CLINICAL TRIAL: NCT01972048
Title: Mobile Phone Multimedia Messaging Intervention for Breast Cancer Screening: Intervention Phase
Brief Title: Mobile Phone Multimedia Messaging Intervention for Breast Cancer Screening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left University
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013NTLS063
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast cancer screening; mammogram
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Participants in the control group will receive the mailed print brochure about breast cancer screening and community resources.
  Interventions: Other: Print brochure
- Intervention group (Experimental): Participants will receive the mMammogram intervention.
  Interventions: Behavioral: mMammogram

INTERVENTIONS:
Behavioral: mMammogram — Text messages delivered via mobile app to participants designed to inform them about breast cancer screening and encourage them to schedule a mammogram.
  Arms: Intervention group
Other: Print brochure — Mailed print brochure about breast cancer screening and community resources.
  Arms: Control group

SUMMARY:
Korean American (KA) women have among the highest breast cancer mortality rates and lowest breast cancer screening rates of U.S. American women across racial/ethical groups. This innovative project seeks to harness mobile phone technology as a means to take preventative health care to a new level among this population. Using the Fogg Behavioral Model this study proposes to develop a mobile phone-based intervention designed to motivate KA women to undergo an annual mammogram (mMammogram). The overall study aim is to develop and assess the feasibility and effectiveness of a 7-day long mMammogram intervention designed to persuade KA women to undergo breast cancer screening.

DETAILED DESCRIPTION:
Specific aims over the three-year period include the following: (1) The first year will be devoted to intervention and protocol development. A major emphasis in year 1 will be developing the community advisory board (CAB), conducting a series of pre-intervention focus groups, and working with pertinent persuasive technology consultants to develop and pilot-test the intervention. (2) The second year and the first half of the third year will focus on delivery of the intervention. (3) the second half of the third year will be devoted to data analysis and dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Korean American immigrant women
* Aged 40-79
* Residence in Minnesota
* Possession of mobile phone with text-message function
* Possession of active email account

Exclusion Criteria:

* Mammogram receipt within the past 2 years

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Mammogram receipt | 1 week
  The receipt of mammogram (or scheduled appointment) will be measured by self-report.

SECONDARY OUTCOMES:
Breast cancer knowledge | 1 week
  Breast cancer knowledge will be measured by means of McCance, Mooney and Smith's ten-item "Breast Cancer Knowledge" test.
Breast cancer health beliefs | 1 week
  Change in health beliefs will be measured using Champion's Health Belief Model scales.
Culture specific attitudes toward breast cancer | 1 week
  Culture-specific attitudes toward breast cancer screening, such as modesty, will be measured utilizing six items from Tang and colleagues and fatalistic attitudes toward breast cancer will be measured by means of three items from Taylor and colleagues.
Participant intent to undergo screening | 1 week
  We will measure participant intent to undergo screening by use of an adapted version of the transtheoretical model.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Y Lee, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Lee H, Ghebre R, Le C, Jang YJ, Sharratt M, Yee D. Mobile Phone Multilevel and Multimedia Messaging Intervention for Breast Cancer Screening: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 Nov 7;5(11):e154. doi: 10.2196/mhealth.7091. PMID 29113961